CLINICAL TRIAL: NCT02688283
Title: Randomized, Controlled, Cross-over Study Comparing The Effect on Glycemic Responses and Subjective Ratings of Satiety of a Snack With or Without Ingredients to Slow Carbohydrate Digestion
Brief Title: The Effect on Glycemic Responses and Subjective Ratings of Satiety of a Snack With or Without Ingredients to Slow Carbohydrate Digestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1512
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Glycemic Response; Satiety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test-cluster (Experimental): 56g of optimized savory cluster made through a proprietary process with slowly digestible carbohydrates and fiber
  Interventions: Other: Nutrient cluster
- Control-cluster (Placebo Comparator): 56g of control cluster made from general baking process with typical ingredients commonly used in commercially available energy snacks or bars
  Interventions: Other: Nutrient cluster
- White-bread (Placebo Comparator): 45g of white bread containing equivalent amount of available carbohydrate in 56g of optimized savory cluster
  Interventions: Other: Nutrient cluster

INTERVENTIONS:
Other: Nutrient cluster — Test cluster is an optimized savory cluster made through a proprietary baking process combined with slow digestible carbohydrates and fiber

SUMMARY:
The objective of this trial is to compare a snack with ingredients (whole grains and dietary fiber) to slow carbohydrate digestion to a similar control snack without such ingredients and evaluate the effect of the snack on glycemic response and subjective satiety. The test product will be compared with a control product as well as white bread in a randomized, controlled, crossover trial including 20 healthy males or females between the ages of 18 and 70 and having a body mass index (BMI) between 25 and 30 kg/m2. Following an overnight fast, participants will be given each of the study products in a random order at least a week apart. Glucose and insulin will be measured before product consumption and over a period of four hours. Visual analog scales to measure subjective satiety will also be administered over a period of four hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between the ages of 18 and 70 inclusive
2. No chronic medications other than oral contraceptives
3. Body Mass Index (BMI) between 25 and 30 kg/m2 inclusive.
4. Body weight stable in a 5 kg range in the 3 months prior to study entry

Exclusion Criteria:

1. Pregnant or nursing a baby
2. Women with child-bearing potential who are unwilling to use an effective means of contraception during the study which could include abstinence.
3. Adults unable to consent and prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) for glucose and insulin | 0-4 hours post consumption

SECONDARY OUTCOMES:
AUC for the visual analog scale (VAS) ratings of satiety | 0-4 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center

IPD SHARING:
Plan to Share IPD: No